CLINICAL TRIAL: NCT04523675
Title: Effects of NAC Supplementation on Immune Function, Inflammatory and Performance Responses of Elite Soccer Players Participated in Three Repetitive Games.
Brief Title: NAC Supplementation and Soccer Specific Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Ioannis G. Fatouros, Associate Professor, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NAC-SOCCER-2016
Record Dates: First submitted 2020-06-22; First posted 2020-08-21 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Skeletal Muscle Damage; Exercise-induced Aseptic Inflammation; Skeletal Muscle Performance; Antioxidant Status
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- EXP-NAC (Experimental): Participated in daily training sessions and three games, and supplemented daily with N-acetylcysteine, orally in three daily dosages (morning-midday-evening),for seven consecutive days.
  Interventions: Dietary Supplement: N-acetylcysteine
- EXP-Pla (Experimental): Participated in daily training sessions and three games, and supplemented daily with Placebo, orally in three daily dosages (morning-midday-evening), for seven consecutive days.
  Interventions: Dietary Supplement: Placebo
- CON-NAC (Active Comparator): Participated in daily training sessions only and supplemented daily with N-acetylcysteine, orally in three daily dosages (morning-midday-evening),for seven consecutive days.
  Interventions: Dietary Supplement: N-acetylcysteine
- CON-Pla (Active Comparator): Participated in daily training sessions only and supplemented daily with Placebo, orally in three daily dosages (morning-midday-evening), for seven consecutive days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: N-acetylcysteine — Orally in three daily dosages (morning-midday-evening), at 20 mg/kg/day, for seven consecutive days.
  Other Names: NAC
  Arms: CON-NAC; EXP-NAC
Dietary Supplement: Placebo — 500 mL drink that contained water (375 mL), sugar-free cordial (125 ml), and 2 g of low-calorie glucose/dextrose powder. Orally in three daily dosages (morning-midday-evening), for seven consecutive days.
  Arms: CON-Pla; EXP-Pla

SUMMARY:
In this investigation the investigators utilized NAC supplementation to boost GSH availability during an one-week-microcycle consisting of three soccer games, in order to test the hypotheses that: i) antioxidant supplementation may enhance the recovery of performance and physiological stress variables following multiple match-plays and ii) redox status perturbations are critical in regulating the inflammatory response and repair in skeletal muscle, following repetitive exercise-induced muscle injuries.

DETAILED DESCRIPTION:
After exercise-induced muscle microtrauma the thiol/disulfide couple of reduced (GSH) and oxidized glutathione (GSSG) is a key regulator of important transcriptional pathways that control the inflammatory response and recovery of skeletal muscle.

The objective was to examine how thiol-based antioxidant supplementation affects the muscle damage, oxidative stress, inflammatory and immune responses, as well as the level of post-game fatigue and muscle's recovery kinetics in response to three soccer games within a week. Participants were randomly assigned to one of four groups: i) Experimental-NAC [EXP-NAC, N=10, participated in daily training sessions and three games and received NAC (20 mg/kg/day)], ii) Experimental-Placebo (EXP-Pla, N=10, participated in daily training sessions and three games and received Placebo), iii) Control-NAC [CON-NAC, N=10, participated in daily training sessions only and received NAC(20 mg/kg/day)] and iv) Control-Placebo (CON-Pla, N=10, participated in daily training sessions only and received Placebo). Blood samples were collected at baseline, post-games and daily during recovery. Performance was assessed at baseline and daily during recovery.

ELIGIBILITY:
Inclusion Criteria:

* Participation at elite level (top three division leagues) of soccer competition for at least five years
* Abstained from consumption of performance-enhancing supplements, antioxidant supplements and medications (for at least 6 months before and during the study)
* Participation in at least six two-hour training sessions and one match per week
* Non-smokers

Exclusion Criteria:

* A known NAC intolerance or allergy
* A recent febrile illness
* History of muscle lesion
* Lower limb trauma
* Metabolic diseases

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in total antioxidant capacity in serum | At baseline and daily throughout the study, up to 11 days
Change in protein carbonyls in serum | At baseline and daily throughout the study, up to 11 days
Change in thiobarbituric acid reactive substances in serum | At baseline and daily throughout the study, up to 11 days
Change in reduced glutathione in red blood cells | At baseline and daily throughout the study, up to 11 days
Change in oxidized glutathione in red blood cells | At baseline and daily throughout the study, up to 11 days
Change in creatine kinase in activity in plasma | At baseline and daily throughout the study, up to 11 days
Change in white blood cell count in blood | At baseline and daily throughout the study, up to 11 days
Change in repeated sprint ability | At baseline and daily throughout the study, up to 11 days
  Players' repeated sprint ability was assessed via a repeared sprint test. Each player performed 5 x 30 meters sprints interspersed by 25 seconds of active recovery. Sprint time was recorded by using infrared photoelectrical gates.
Change in high intensity running during the game | During games 1, 2 and 3
  High intensity running (i.e. > 14km/h) during the games was monitored by utilizing high time-resolution GPS devices.

SECONDARY OUTCOMES:
Change in blood lactate concentration during the game | During games 1, 2 and 3
Change in average heart rate during the game | During games 1, 2 and 3

CONTACTS AND LOCATIONS:
Overall Officials: IOANNIS G FATOUROS, Ph.D., Principal Investigator — UNIVERSITY OF THESSALY, SCHOOL OF PHYSICAL EDUCATION & SPORTS SCIENCES
Locations (1):
- Exercise Biochemistry Laboratory, School of Physical Education & Sports Sciences, University of Thessaly, Trikala, Greece